CLINICAL TRIAL: NCT01696474
Title: Short Course of Bortezomib in Anemic Patients With Refractory Cold Agglutinin Disease
Acronym: CAD0111
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAD0111; EudraCT number 2011-006329-42
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Refractory Cold Agglutinin Disease
Keywords: Refractory cold agglutinin disease; Bortezomib; blood-transfusion
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib therapy (Experimental): A single course of Bortezomib will be given at the dose of 1,3 mg/sqm iv on days 1, 4, 8, 11. Prophylaxis of HZ reactivation will be given with oral acyclovir at the dosage of 400 mg twice daily for one month after the end of Bortezomib.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
This multicenter, phase II, open label study will enroll patients with chronic cold agglutinin disorder. A single course of Bortezomib will be given at the dose of 1,3 mg/sqm iv on days 1, 4, 8, 11.

DETAILED DESCRIPTION:
Based on its activity in MM, single agent Bortezomib was tested in phase II trials in lymphoplasmacytic lymphoma, the disorder most frequently associated with CAD, and achieved 40-80% responses. These striking clinical responses indicate that proteasome activity is critical for the survival of immunoglobulin-secreting cells. The resolution of transfusion requirement in two patients with refractory CAD associated with IgMk monoclonal gammopathy has been reported after treatment with a short course of Bortezomib. It may be interesting to test the efficacy of Bortezomib in a larger series of patients with refractory CAD, idiopathic or associated with an otherwise asymptomatic B cell clonal disorder, and to evaluate the duration of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic cold agglutinin disorder requiring or with a hemoglobin concentration below 10g/L determined at least monthly during the two months before entering the trial;
* Failure of at least one previous treatment attempt;
* Hemoglobin level assessment;
* Presence of serum cold agglutinin (CA). If an overnight incubation is used for CA detection, a titer at 4°C of 64 or higher is required;
* Written informed consent.

Exclusion Criteria:

* Presence of a concomitant lymphoproliferative disorder requiring specific treatment for reasons other than cold agglutinin related hemolytic anemia;
* Preexisting peripheral neuropathy;
* Known hypersensitivity to Bortezomib;
* Non-cooperative behaviour or non-compliance;
* Psychiatric diseases or conditions that might impair the ability to give informed consent;
* Patients who are pregnant (women of childbearing potential must have a negative serum pregnancy test). Post-menopausal women must be amenorrhoic for at least 24 months to be considered of non-childbearing potential. Male and female patients must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-12; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
Number of patients who become transfusion-free after Bortezomib therapy. | After 3 months from study entry.
  Cumulative proportion of patients transfusion-free at three months after Bortezomib therapy.
Number of patients who have never been transfused with a >2g hemoglobin rise compared to baseline. | After 3 months from study entry.

SECONDARY OUTCOMES:
Number of CTC grade 3 and 4 adverse events. | After 12 months from study entry.
  Evaluation of the incidence of CTC grade 3 and 4 adverse events during and after treatment.
Duration in months of transfusion independence. | At 12 months from study entry.
Effect of treatment on the underlying clonal B cell disorder. | At 3 months from study entry.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Rossi, Dr., Principal Investigator — S.C. Ematologia e Dipartimento di Oncologia Medica Spedali Civili - Brescia
Locations (8):
- Italy (8):
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Centro Trapianti di Midollo - IRCCS Ospedale Maggiore Policlinico, Milan
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - U.O. Ematologia Clinica - Azienda USL di Pescara, Pescara
  - Azienda Ospedaliera Bianchi Melacrino Morelli, Reggio Calabria
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Ospedale San Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No